CLINICAL TRIAL: NCT06618950
Title: The Effect of Physical Activity on Healthy Lifestyle, Self-Esteem and Psychological Well-Being in Late Adolescents: A Randomized Controlled Study
Brief Title: The Effects of Physical Activity on Healthy Lifestyle, Self-Esteem and Psychological Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hakan Avan, doktor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: hakanavan-0002
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Physical Activity Awareness; Healthy Lifestyle Behaviors
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: physical activity — The key factor that distinguishes this study from others is its comprehensive examination of the effects of regular physical activity on late adolescents, not only in terms of physical health but also regarding healthy lifestyle behaviors, self-esteem, and psychological well-being. While other studies typically focus on the benefits of physical activity for physical health, this research considers the broader psychological and social development of adolescents, offering a wider perspective. Additionally, its emphasis on the sustainability of a planned and structured physical activity regimen, along with its approach to transforming physical activity into a lifestyle, represents a significant difference.
  Arms: Intervention

SUMMARY:
Introduction Adolescence is a critical developmental stage marked by significant physical, emotional, cognitive, and social changes. Establishing healthy lifestyle habits during this time is essential for overall well-being.

Health Promotion Health promotion enhances individual well-being through self-regulation and the adoption of healthy behaviors, including physical activity, proper nutrition, safe sexual practices, stress management, and avoidance of harmful substances.

Importance of Physical Activity Physical activity tends to decline in adolescence but is vital for mental health, reducing anxiety and depression, and boosting self-esteem and academic performance.

Planning Physical Activity Engaging in regular, planned physical activity is crucial for maintaining its benefits. Inconsistent participation can lead to diminished positive effects.

Research Objective This study investigates the impact of regular physical activity on the healthy lifestyle behaviors, self-esteem, and psychological well-being of late adolescents.

Research Hypotheses

1. Physical activity positively affects healthy lifestyle behaviors.
2. Physical activity enhances self-esteem.
3. Physical activity improves psychological well-being. Method An analytical interventional study will involve students aged 18-21 from Kahramanmaraş Sutcu Imam University. Participants will be randomly assigned to either an intervention group (12-week physical activity program) or a control group (routine education). Both groups will complete pre- and post-tests using established scales.

Inclusion/Exclusion Criteria Participants must be students aged 18-21, willing to participate, and complete the study without missing sessions. Incomplete questionnaires will lead to exclusion.

Statistical Analysis A total of 84 participants will be involved. Descriptive and inferential statistical analyses will be conducted using SPSS, with significance set at p < 0.05.

This study aims to clarify how regular physical activity influences the health and well-being of adolescents, contributing to healthier lifestyle choices.

DETAILED DESCRIPTION:
Introduction The adolescent period is the phase of life characterized by the fastest growth and development, marking the transition from childhood to adulthood. During this time, adolescents experience a sensitive period in which they complete their physical, emotional, cognitive, sociocultural, vocational, and moral development. It is crucial to establish healthy lifestyle behaviors during adolescence and to promote adolescent health for a healthy society.

Health Promotion Health promotion is defined as the increase in the well-being of an individual or group and the realization of one's potential This process can be achieved in adolescents through self-regulation and transforming healthy lifestyle behaviors into permanent habits. Healthy lifestyle behaviors include engaging in physical activity, maintaining a healthy diet, practicing safe sexual behaviors, managing stress, and avoiding harmful habits such as smoking, alcohol, and substance use.

Importance of Physical Activity Physical activity among adolescents noticeably declines compared to earlier stages and continues to decrease with age into adulthood. Physical activity has been shown to be an effective way to enhance mental health and well-being. Individuals who are physically active exhibit lower levels of fatigue, anxiety, stress, and depression, along with greater vitality and well-being during both adolescence and adulthood.

Adolescents who engage in physical activity tend to have an ideal body weight and shape, exhibit more cheerful and positive peer interactions, achieve higher academic success, and demonstrate greater responsibility and independent decision-making skills. Their self-confidence and self-esteem significantly increase during this process Planning Physical Activity Adolescents can perform physical activities that are appropriate for their age group and of their choosing in their daily lives. However, it is important to remember that the chosen activity should be planned, regular, continuous, and of appropriate intensity. Otherwise, the positive effects of physical activity may not be realized and may not become permanent. When physical activity does not transition into a regular and planned program, or when the activity is abandoned, the beneficial effects can quickly diminish.

The key factor that distinguishes this study from others is its comprehensive examination of the effects of regular physical activity on late adolescents, not only in terms of physical health but also regarding healthy lifestyle behaviors, self-esteem, and psychological well-being. While other studies typically focus on the benefits of physical activity for physical health, this research considers the broader psychological and social development of adolescents, offering a wider perspective. Additionally, its emphasis on the sustainability of a planned and structured physical activity regimen, along with its approach to transforming physical activity into a lifestyle, represents a significant difference.

Research Objective This study aims to determine the effects of regular physical activity on the healthy lifestyle behaviors, self-esteem, and psychological well-being of late adolescents. In this context, the goal is to better understand the impact of regular physical activity on adolescent health.

Research Hypotheses H1: Does physical activity have an effect on healthy lifestyle behaviors? H2: Does physical activity have an effect on self-esteem? H3: Does physical activity have an effect on psychological well-being? Method This study, planned as an analytical interventional research, will focus on students aged 18-21 from the Kahramanmaraş Sutcu Imam University School of Health Services. Individuals who voluntarily participate, meet the specified criteria, and answer the questionnaire will constitute the sample of the study. A simple random sampling method will be used for the sample selection.

Research Flow The research will be conducted between 13 October 2024 and 03 January 2025. Expert opinions will be obtained for educational materials and physical activity methods. Institutional permission will be secured, and an informed consent form will be distributed to the students. Participants who volunteer for the study will be assigned numbers, and intervention and control group participants will be determined using simple random sampling. Gender, age, and BMI (Body Mass Index) will be used as randomization criteria for the intervention and control groups. Both groups will undergo a pre-test.

Participants in the control group will continue their routine education, while participants in the intervention group will first receive training on physical activity and its benefits, followed by an 12-week physical activity program. For the intervention group, the first three weeks will involve moderate-intensity brisk walking and light jogging twice a week for 15-30 minutes, followed by brisk walking and moderate jogging twice a week for 30 minutes in weeks 4, 5 and 6. In the last six weeks, the activities will include brisk walking and high-intensity jogging twice a week for 30-45 minutes. At the end of the twelve weeks, both the intervention and control groups will undergo a post-test.

Inclusion Criteria for Participants Must be a student at Kahramanmaraş Sutcu Imam University School of Health Services, Aged between 18-21, Must be willing to participate in the research. Exclusion Criteria for Participants Incomplete questionnaire forms, Failure to participate in at least one physical activity session. Measured Variables Dependent Variables: Scores from the Healthy Lifestyle Behaviors Scale, Self-Esteem Scale, and Psychological Well-Being Scale.

Independent Variables: Socio-demographic questions. Statistical Analysis of the Research Sample Size Calculation Method: Based on the power analysis conducted on students aged 18-21 who are willing to participate in the study (two-tailed hypothesis, 5% error margin, 95% power, 0.8 effect size), a total of 84 participants (42 control, 42 intervention) will constitute the sample of the study.

Descriptive Statistical Measures: Count, percentage, mean, standard deviation. Normality Test and/or Homogeneity of Variance Test: The normality of the data will be evaluated using Skewness and Kurtosis (±1) values and the Shapiro-Wilk normality test. Homogeneity of variances will be assessed using Levene's test.

Comparison Groups and Analytical Statistical Methods: Data will be analyzed using IBM SPSS Statistics Standard Concurrent User V 26 (IBM Corp., Armonk, New York, USA). The normal distribution of numerical variables will be tested with the Shapiro-Wilk normality test. Homogeneity of variances will be evaluated using Levene's test. Independent samples t-test will be used for comparing BMI values between groups. Fisher's exact test will be used for comparing categorical variables between groups. Pre-test and post-test scale scores will be compared using two-way ANOVA for repeated measures. Bonferroni correction will be applied for the comparison of main effects in ANOVA. A p-value of <0.05 will be considered statistically significant. The content validity testing of educational materials will be conducted using the Lawshe method.

Potential Outcomes of This Study:

Physical Activity and Healthy Lifestyle:

* Regular physical activity among late adolescents may enhance healthy lifestyle behaviors.
* A positive relationship between physical activity and healthy eating habits and other healthy behaviors.

Self-Esteem:

* Evidence suggesting that regular physical activity increases self-esteem.
* Physical activity may positively influence adolescents' self-confidence and social interactions.

Psychological Well-Being:

* Data indicating that physical activity is effective in reducing levels of anxiety, stress, and depression.
* A conclusion that increases in psychological well-being are linked to physical activity.

Psychological Well-Being:

* Physical activity may positively impact adolescents' social skills and peer relationships.
* The encouraging effects of regular physical activity on group interaction and teamwork.

Long-Term Health Benefits:

* The potential for regular physical activity to transform into lasting health behaviors beyond adolescence.
* Habits acquired during late adolescence may contribute to sustainable health behaviors in adulthood.

Education and Intervention Programs:

* The necessity for developing educational and intervention programs that promote physical activity based on the study's findings.
* Recommendations for strategies to increase physical activity at school and community levels.

Emotional Regulation:

The potential of regular physical activity to enhance emotional regulation skills.

ELIGIBILITY:
Inclusion Criteria:

* Must be a student at Kahramanmaraş Sutcu Imam University School of Health Services,
* Aged between 18-21,
* Must be willing to participate in the research.

Exclusion Criteria:

* Incomplete questionnaire forms,
* Failure to participate in at least one physical activity session.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-10-13 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Development of Healthy Lifestyle behaviors | 12 weeks
  Health promotion can be achieved by transforming self-regulation and healthy lifestyle behaviors into permanent habits in adolescents. For this purpose, the Healthy Lifestyle Behaviors Scale will be used. The Healthy Lifestyle Behaviors Scale allows the determination of healthy lifestyle behaviors at all stages of adolescence. The maximum score that can be obtained from the scale is 160 and the minimum score is 40. Although there is no cut-off point, it is reported that as the score increases, the level of positive health behaviors also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Eyalet/Yerleşke, Turkey (Türkiye)